CLINICAL TRIAL: NCT06491173
Title: Assessment of Accuracy, Precision, and Feasibility of a Handheld Near-Infrared Light Device (InfraScanner 2500™) in Detecting Traumatic Intracranial Hemorrhage in Uganda
Brief Title: Detecting Traumatic Intracranial Hemorrhage With the InfraScanner 2500™ in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Mbarara Regional Referral Hospital (Unknown); Mayanja Memorial Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00115721
Record Dates: First submitted 2024-07-01; First posted 2024-07-08 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-08

CONDITIONS: Head Trauma; Crushing Skull Injury; Head Injury; Head Injuries, Multiple; Head Injuries, Closed; Head Trauma,Closed; Head Injury Major; Head Injury, Minor; Head Injury, Open; Injury, Craniocerebral; Injury, Head; Multiple Head Injury; Trauma, Head; Head Trauma Injury; Head Trauma, Penetrating; Craniocerebral Injury
MeSH Terms: conditions — Craniocerebral Trauma; Head Injuries, Closed; Head Injuries, Penetrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- InfraScanner 2500™ (Experimental): All patients entered into the trial will undergo at least one cranial scanning using the InfraScanner 2500™ upon arrival to the casualty unit at MRRH following CT. Patients will be scanned using the InfraScanner 2500™ following each subsequent CT as allowed by patient or representative. Patients will know the results of the CT but not the InfraScanner 2500™. The standard for comparison will be determined as follows. A CT result that is positive for hematoma will be considered a true positive and a CT result that is negative for hematoma will be considered a true negative. In cases where the results of the CT are negative for hematoma and the results of the InfraScanner 2500™ are positive consideration of further follow-up will be given on a case-by-case basis.
  Interventions: Device: InfraScanner 2500™

INTERVENTIONS:
Device: InfraScanner 2500™ — The Infrascanner is a portable screening device that uses Near-Infrared (NIR) technology to screen patients for intracranial bleeding, identifying those who would most benefit from immediate referral to a CT scan and neurosurgical intervention.

SUMMARY:
The goal of this study is to determine the sensitivity, specificity, and positive and negative predictive values of the portable near-infrared-based device (portable NIR-based device), the InfraScanner 2500™, to detect intracranial hematomas (epidural hematomas (EDH) and/or subdural hematomas (SDH)) in patients hospitalized at Mbarara Regional Referral Hospital (MRRH) or Mayanja Memorial Hospital (MMH) who have sustained or who are suspected to have sustained head trauma.

DETAILED DESCRIPTION:
When applicable (conscious patient and/or family or legally authorized representative is present) the study will be introduced to the patient and relevant parties prior to the research team approaching the patient. While head trauma frequently results in impaired cognition and/or consciousness, and due to the urgency of these circumstances patients are often not accompanied by kin, whenever appropriate, the purpose of the research and the procedure will be explained in detail with all questions answered to the patient's and/or representative's satisfaction. Because patients who sustain head trauma injuries typically remain within the hospital for multiple days for monitoring and care, each participant may undergo multiple Computed Tomography (CT) scans over the course of his or her hospitalization, affording the opportunity of one to numerous measurements from each patient during his or her hospital stay.

Upon presentation to the casualty unit at MRRH or MMH and following each CT scan, the study team will approach the patient to scan the patient's cranium with the InfraScanner 2500™. If permission is granted, the study team member sequentially measures the optical absorption for each of the 8 quadrants of the scalp (frontal, temporal, parietal, and occipital bilaterally). The device is engineered such that the light emitter and receiver are spaced 4 cm apart, allowing the light's intensity to be measured between adjacent light guides. This entire procedure, including greeting and scanning the patient should take <10 minutes. Subsequent CT scan(s) the patient receives determines the number of potential data collections.

The patient and/or representative may refuse a scan during any encounter, and as such, the scan will not be done. For each patient scanned with the InfraScanner 2500™ they will be de-identified with a subject number, with age, sex, gender, skin color, hair color, hair thickness, mechanism of injury, Glasgow Coma Scale score, and mean time elapsed between CT scan and near-infrared measurement. These data will be stored in de-identified form on the Research Electronic Data Capture (REDCap) database and/or Microsoft Excel on a secured network drive within the Department of Neurosurgery at Duke.

The collection period for each research subject concludes 30-days following his or her initial measurement with the InfraScanner 2500™, patient discharge, or patient death.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who presents to MRRH or MMH with suspected head trauma, who is able to, or who has a legally authorized representative who is able to consent in English, Swahili, or Luganda will be considered for this study.

Exclusion Criteria:

* Patients for which wounds to their head are too large to properly use the InfraScanner 2500™ will be excluded from this study. Patients will also be excluded if hair cannot be appropriately parted to allow for the fiberoptic tips of the device to make direct contact with the scalp. Patients for whom it is not possible to obtain an Infrascan within 30 minutes of their CT imaging will also be excluded from the study.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Detection of Intracranial hemorrhage (ICH) by the InfraScanner 2500™ Stratified by CT Positive and CT Negative Status | Within 30 minutes following CT scan
  Precision of the InfraScanner 2500™ relative to CT scans in an African, LMIC (lower middle income country) population.

SECONDARY OUTCOMES:
Number of Participants With Detection of Intracranial hemorrhage (ICH) by the InfraScanner 2500™ | Within 30 minutes following CT scan
  Accuracy of the InfraScanner 2500™ in darker-skinned populations within LMICs.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kolls, MD, PhD, Principal Investigator — Duke University
Locations (2):
- Uganda (2):
  - Mayanja Memorial Hospital, Mbarara
  - Mbarara Regional Referral Hospital, Mbarara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dewan MC, Rattani A, Gupta S, Baticulon RE, Hung YC, Punchak M, Agrawal A, Adeleye AO, Shrime MG, Rubiano AM, Rosenfeld JV, Park KB. Estimating the global incidence of traumatic brain injury. J Neurosurg. 2018 Apr 27;130(4):1080-1097. doi: 10.3171/2017.10.JNS17352. Print 2019 Apr 1. PMID 29701556
- [Background] Veerappan VR, Gabriel PJ, Shlobin NA, Marks K, Ooi SZY, Aukrust CG, Ham E, Abdi H, Negida A, Park KB, El Ouahabi A. Global Neurosurgery in the Context of Global Public Health Practice-A Literature Review of Case Studies. World Neurosurg. 2022 Sep;165:20-26. doi: 10.1016/j.wneu.2022.06.022. Epub 2022 Jun 11. PMID 35697226
- [Background] Ukachukwu AK, Still MEH, Seas A, von Isenburg M, Fieggen G, Malomo AO, Shokunbi MT, Egger JR, Haglund MM, Fuller AT. Fulfilling the specialist neurosurgical workforce needs in Africa: a systematic review and projection toward 2030. J Neurosurg. 2022 Aug 12;138(4):1102-1113. doi: 10.3171/2022.2.JNS211984. Print 2023 Apr 1. PMID 35962968
- [Background] Janca A, Aarli JA, Prilipko L, Dua T, Saxena S, Saraceno B. WHO/WFN Survey of neurological services: a worldwide perspective. J Neurol Sci. 2006 Aug 15;247(1):29-34. doi: 10.1016/j.jns.2006.03.003. Epub 2006 Apr 19. PMID 16624322
- [Background] Ttendo SS, Was A, Preston MA, Munyarugero E, Kerry VB, Firth PG. Retrospective Descriptive Study of an Intensive Care Unit at a Ugandan Regional Referral Hospital. World J Surg. 2016 Dec;40(12):2847-2856. doi: 10.1007/s00268-016-3644-5. PMID 27506722
- [Background] Vaca SD, Feng AY, Ku S, Jin MC, Kakusa BW, Ho AL, Zhang M, Fuller A, Haglund MM, Grant G. Boda Bodas and Road Traffic Injuries in Uganda: An Overview of Traffic Safety Trends from 2009 to 2017. Int J Environ Res Public Health. 2020 Mar 22;17(6):2110. doi: 10.3390/ijerph17062110. PMID 32235768
- [Background] Firth PG, Mushagara R, Musinguzi N, Liu C, Boatin AA, Mugabi W, Kayaga D, Naturinda P, Twesigye D, Sanyu F, Mugyenyi G, Ngonzi J, Ttendo SS; Mbarara SQUAD Consortium. Surgical, Obstetric, and Anesthetic Mortality Measurement at a Ugandan Secondary Referral Hospital. Anesth Analg. 2021 Dec 1;133(6):1608-1616. doi: 10.1213/ANE.0000000000005734. PMID 34415855
- [Background] Hyam JA, Welch CA, Harrison DA, Menon DK. Case mix, outcomes and comparison of risk prediction models for admissions to adult, general and specialist critical care units for head injury: a secondary analysis of the ICNARC Case Mix Programme Database. Crit Care. 2006;10 Suppl 2(Suppl 2):S2. doi: 10.1186/cc5066. PMID 17352796
- [Background] Nigatu AM, Yilma TM, Gezie LD, Gebrewold Y, Gullslett MK, Mengiste SA, Tilahun B. Medical imaging consultation practices and challenges at public hospitals in the Amhara regional state, Northwest Ethiopia: a descriptive phenomenological study. BMC Health Serv Res. 2023 Jul 24;23(1):787. doi: 10.1186/s12913-023-09652-9. PMID 37488569
- [Background] Feiner JR, Severinghaus JW, Bickler PE. Dark skin decreases the accuracy of pulse oximeters at low oxygen saturation: the effects of oximeter probe type and gender. Anesth Analg. 2007 Dec;105(6 Suppl):S18-S23. doi: 10.1213/01.ane.0000285988.35174.d9. PMID 18048893
- [Background] Gottlieb ER, Ziegler J, Morley K, Rush B, Celi LA. Assessment of Racial and Ethnic Differences in Oxygen Supplementation Among Patients in the Intensive Care Unit. JAMA Intern Med. 2022 Aug 1;182(8):849-858. doi: 10.1001/jamainternmed.2022.2587. PMID 35816344
- [Background] Valbuena VSM, Seelye S, Sjoding MW, Valley TS, Dickson RP, Gay SE, Claar D, Prescott HC, Iwashyna TJ. Racial bias and reproducibility in pulse oximetry among medical and surgical inpatients in general care in the Veterans Health Administration 2013-19: multicenter, retrospective cohort study. BMJ. 2022 Jul 6;378:e069775. doi: 10.1136/bmj-2021-069775. PMID 35793817
- [Background] Ries AL, Prewitt LM, Johnson JJ. Skin color and ear oximetry. Chest. 1989 Aug;96(2):287-90. doi: 10.1378/chest.96.2.287. PMID 2752811
- [Background] Okunlola OE, Lipnick MS, Batchelder PB, Bernstein M, Feiner JR, Bickler PE. Pulse Oximeter Performance, Racial Inequity, and the Work Ahead. Respir Care. 2022 Feb;67(2):252-257. doi: 10.4187/respcare.09795. Epub 2021 Nov 12. PMID 34772785
- [Background] Jamali H, Castillo LT, Morgan CC, Coult J, Muhammad JL, Osobamiro OO, Parsons EC, Adamson R. Racial Disparity in Oxygen Saturation Measurements by Pulse Oximetry: Evidence and Implications. Ann Am Thorac Soc. 2022 Dec;19(12):1951-1964. doi: 10.1513/AnnalsATS.202203-270CME. PMID 36166259
- [Background] Braun T, Kunz U, Schulz C, Lieber A, Willy C. [Near-infrared spectroscopy for the detection of traumatic intracranial hemorrhage: Feasibility study in a German army field hospital in Afghanistan]. Unfallchirurg. 2015 Aug;118(8):693-700. doi: 10.1007/s00113-013-2549-0. German. PMID 24435101
- [Background] Albutt K, Punchak M, Kayima P, Namanya DB, Anderson GA, Shrime MG. Access to Safe, Timely, and Affordable Surgical Care in Uganda: A Stratified Randomized Evaluation of Nationwide Public Sector Surgical Capacity and Core Surgical Indicators. World J Surg. 2018 Aug;42(8):2303-2313. doi: 10.1007/s00268-018-4485-1. PMID 29368021
- [Background] Atumanya P, Sendagire C, Wabule A, Mukisa J, Ssemogerere L, Kwizera A, Agaba PK. Assessment of the current capacity of intensive care units in Uganda; A descriptive study. J Crit Care. 2020 Feb;55:95-99. doi: 10.1016/j.jcrc.2019.10.019. Epub 2019 Nov 4. PMID 31715537
- [Background] Koltai DC, Dunn TW, Smith PJ, Sinha DD, Bobholz S, Kaddumukasa M, Kakooza-Mwesige A, Kajumba M, Smith CE, Kaddumukasa MN, Teuwen DE, Nakasujja N, Chakraborty P, Kolls BJ, Nakku J, Haglund MM, Fuller AT. Sociocultural determinants and patterns of healthcare utilization for epilepsy care in Uganda. Epilepsy Behav. 2021 Jan;114(Pt B):107304. doi: 10.1016/j.yebeh.2020.107304. Epub 2020 Aug 4. PMID 32768344
- [Background] Buderer NM. Statistical methodology: I. Incorporating the prevalence of disease into the sample size calculation for sensitivity and specificity. Acad Emerg Med. 1996 Sep;3(9):895-900. doi: 10.1111/j.1553-2712.1996.tb03538.x. PMID 8870764
- [Background] Robertson CS, Zager EL, Narayan RK, Handly N, Sharma A, Hanley DF, Garza H, Maloney-Wilensky E, Plaum JM, Koenig CH, Johnson A, Morgan T. Clinical evaluation of a portable near-infrared device for detection of traumatic intracranial hematomas. J Neurotrauma. 2010 Sep;27(9):1597-604. doi: 10.1089/neu.2010.1340. PMID 20568959
- See also: InfraScan. Infrascanner - White Paper A Handheld Brain Hematoma Detector. Accessed February 4, 2024. — http://infrascanner.com/wp-content/uploads/2018/11/Infrascanner-white-paper-02.18.pdf
- See also: Sample size calculator . Published online 2024. — http://wnarifin.github.io